CLINICAL TRIAL: NCT05216575
Title: Use of Almitrine in COVID-19 Patients With Acute Respiratory Distress Syndrome Treated by High-flow Nasal Canula Oxygen Therapy
Brief Title: Almitrine in COVID-19 Patients With ARDS Treated by HFNO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22reamedcovid01
Record Dates: First submitted 2022-01-28; First posted 2022-01-31 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: ARDS; Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Almitrine treated patients: Administration of Almitrine in spontaneoulsy breathing COVID-19 patients with moderate to severe ARDS treated by high-flow nasal canula oxygen therapy as first-line ventilatory support with persitent severe hypoxemia after awake prone positioning.
  Interventions: Drug: Administration of Almitrine

INTERVENTIONS:
Drug: Administration of Almitrine — Administration of Almitrine (intravenous bolus of 0.5 mg/kg over 30 minutes followed by a continuous perfusion of 16 mg/kg/min in responders)

SUMMARY:
The purpose of this study is to determine the effects of Almitrine administration on oxygenation in COVID-19 patients with acute respiratory distress syndrome treated by high-flow nasal canula oxygen therapy as first-line ventilatory support.

DETAILED DESCRIPTION:
From December 2019, the emergent coronavirus SARSCoV-2 is responsible for the worldwide pandemic of coronavirus disease (COVID-19). Although SARSCoV-2 infection is mainly responsible for mild respiratory symptoms, up to 70% of hospitalized patients with COVID-19-related pneumoniae may develop severe respiratory disease, progressing to acute respiratory distress syndrome (ARDS). These patients may experience severe but well-tolerated hypoxemia, so-called "happy hypoxemia" which may be related to blunted hypoxic vasoconstriction. Almitrine is a selective pulmonary vasoconstrictor that has been reported to improve the oxygenation in ARDS patients by increasing hypoxic pulmonary vasoconstriction. Some small case series reported that the use of Almitrine in mechanically ventilated COVID-19 patients with ARDS improved oxygenation. Given the "happy hypoxemia" phenomenon, it has been suggested to use high-flow nasal canula therapy (HFNO) as first-line ventilatory support in COVID-19 patients with ARDS, since the risk of aerosolization with HFNO was similar to that with standard oxygen therapy and lower to that with non-invasive ventilation. However, the effects of Almitrine in spontaneously breathing patients with ARDS has not been reported so far. Thus, the main goal of this study is to investigate the effects of Almitrine on oxygenation of COVID-19 patients with ARDS treated by HFNO as first-line ventilatory support. The second goal of this study is to determine the effects of Almitrine on respiratory mechanics and hymodynamics.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated by high-flow nasal canula oxygen
2. Positive COVID-19 real-time reverse transcriptase-polymerase chain reaction assay in nasal swabs
3. Persistent severe hypoxemia after awake prone positioning defined by one or more of the following criteria:

   1. SpO2 < 96% with FiO2 > 80%
   2. PaO2/FiO2 ratio < 100 with FiO2 > 80%
4. Patients treated by Almitrine

Exclusion Criteria:

1. Age <18 years old and pregnant women
2. Patients under legal protection
3. Patients with a do not intubate or do not resuscitate decision
4. Patients requiring immediate invasive mechanical ventilation
5. Contraindication to Almitrine
6. Poor echogenicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are spontaneously breathing COVID-19 patients with moderate to severe ARDS treated by high-flow nasal canula oxygen therapy as first-line ventilatory support with persitent severe hypoxemia after awake prone positioning.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Almitrine-induced increase in Pa02/FiO2 ratio. | The 30-minute duration of Almitrine bolus
  The PaO2/FiO2 ratio will be calculated before and after the bolus of Almitrine. Patients with increase in PaO2/FiO2 ratio > 20% will be considered as responders.

SECONDARY OUTCOMES:
Proportion of patients requiring intubation | ICU stay
  To assess the proportion of patients who will require to be intubated during their ICU stay.
Proportion of patients exhibiting right ventricular failure and/or right ventricular dilation and/or acute core pulmonale after administration of Almitrine. | The 30-minute duration of Almitrine bolus
  To assess the proportion of patients who will experience right ventricular failure and/or right ventricular dilation and/or acute core pulmonale after administration of Almitrine.
Clinical prediction of Almitrine effects | The 30-minute duration of Almitrine bolus
  To test the ability of different respiratory variables and radiological patterns to predict the response to Almitrine in terms of oxygenation
Radiological prediction of Almitrine effects | The 30-minute duration of Almitrine bolus
  To test the ability of different radiological patterns to predict the response to Almitrine in terms of oxygenation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, France

IPD SHARING:
Plan to Share IPD: No
No data sharing plan is scheduled